CLINICAL TRIAL: NCT00482417
Title: Efficacy and Safety Study of MK0359 in Patients With Arthritis (0359-017)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0359-017; 2007_573
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

INTERVENTIONS:
Drug: MK0359

SUMMARY:
Efficacy and Safety Study of MK0359 in Patients with Arthritis

ELIGIBILITY:
Inclusion Criteria:

* You are 18-65 years of age and have Rheumatoid Arthritis
* You must be able to read and understand patient questionnaires

Exclusion Criteria:

* You have had certain types of surgery, certain types of cancer or history of Tuberculosis (TB) or HIV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2002-12; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC